CLINICAL TRIAL: NCT06605001
Title: Delay of Gratification: Life Habits of Delaying and Cascading Effects on Life Outcomes
Brief Title: Development, Attention, and Inhibition Study
Acronym: DAISY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1518244; R01HD086184 (NIH)
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Delaying
Keywords: Delay of Gratification; Waiting; Habits; Academic Outcomes
MeSH Terms: conditions — Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delay of Gratification - Treat (Experimental): Reward presented is a sweet treat.
  Interventions: Other: Delay of Gratification
- Delay of Gratification - Gift (Experimental): Reward presented is a wrapped gift.
  Interventions: Other: Delay of Gratification

INTERVENTIONS:
Other: Delay of Gratification — Children will complete a delay of gratification task with 1 of 2 rewards

SUMMARY:
The goal of this clinical trial is to test the associations of young children's early life experiences with delaying behaviors and links with later life outcomes. The main questions it aims to answer are:

* Do experiences with waiting in early childhood predict delaying behavior in context-specific ways?
* Are links between delaying behavior and life outcomes impacted by social conventions, effort and choices around delaying, or other behaviors?

Participants will:

* Complete two delaying tasks with either a sweet or wrapped gift
* Complete three "Simon says"-like games that measure inhibition, cognitive flexibility and proactive control
* Answer a set of questions about academic readiness
* Answer a set of questions about social conventions
* Complete a waiting game on the computer while a camera records eye movements
* Parents will answer questions about their child's behaviors and experiences at home
* Participants will return after 1 year to repeat a subset of these measures

DETAILED DESCRIPTION:
In sessions 1 and 2, 4-6-year-olds will complete a delay of gratification task (randomly assigned to one of two groups, to delay with either a sweet or a wrapped gift), the NASA Load Index to report perceived demand and effort for the delay of gratification task, a computerized delay choice measure (while pupillometric data is collected), a Go/No-Go task, the NIH Toolbox Dimensional Change Card Sort, a Track-It task, a task measuring sensitivity to social conventions, and Woodcock-Johnson IV Tests of Achievement. Parents will complete the Child Behavioral Checklist (CBCL), the Child Behavior Questionnaire (CBQ), the REEF executive function questionnaire, and questionnaires about demographics and children's experiences waiting at mealtimes, when opening gifts, and in other contexts.

In session 3 (1 year after sessions 1 and 2), participants and parents will repeat the measures from sessions 1 and 2.

ELIGIBILITY:
Typically developing children will be recruited. Participants will be pre-screened for developmental disorders.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Choice Delay | Immediately after and 1 year after intervention
  Pattern of waiting behavior represented by area under the curve (AUC) for wait times.
Executive Functions | Pre-intervention and 1 year after intervention
  Composite scores from the REEF, a questionnaire measuring executive functioning.
Social Conventions | Immediately after and 1 year after intervention
  Social task measuring adherence to social conventions.
Academic Readiness | Immediately after and 1 year after intervention
  Woodcock-Johnson IV Tests of Achievement: Letter-Word Identification and Applied Problems standardized scores.
Inhibitory Control (Go/No-Go) | Immediately after and 1 year after intervention
  Accuracy (No-Go trials) during the Go/No-Go inhibitory control task.
Experiences Waiting at Home | Pre-intervention and 1 year after intervention
  Composite score from a questionnaire developed for this study, measuring experiences with waiting.
Cognitive Flexibility (DCCS) | Immediately after intervention and 1 year after intervention
  Accuracy (perseveration errors) during the Dimensional Change Card Sort (DCCS) task.
Problem Behaviors | Pre-intervention and 1 year after intervention
  Composite and sub-scale scores from CBCL, a questionnaire measuring children&amp;#39;s problem behaviors.

SECONDARY OUTCOMES:
Pupil dilation during delayed choice | Immediately after and 1 year after intervention
  Pupil dilation while waiting for expected reward, or skipping for a new trial.
Behavior while delaying | During initial and 1 year follow-up intervention
  Video coding of targeted behaviors (i.e., anticipatory behavior) during delay of gratification.
Subjective Effort | During initial and 1 year follow-up intervention
  Self-reported demand and effort during the delay of gratification task on the NASA Task Load index.
Proactive Control | During initial and 1 year follow-up intervention
  Accuracy during the Track-It proactive control task.
Child Temperment | Pre-intervention and 1 year after intervention
  Composite score from the CBQ, a questionnaire measuring child temperament.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Mind and Brain, Davis, California, United States